Statistical Analysis Plan Version 1.1 -J2G-MC-JZJQ

An Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food and a Proton Pump Inhibitor on the Single-Dose Pharmacokinetics of LOXO-292 in Healthy Adult Subjects

NCT05468164

Approval Date: 06-Sep-2018



- 16.1.9 Documentation of Statistical Methods
- 16.1.9.1 Statistical Analysis Plan

# Statistical Analysis Plan

An Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food and a Proton Pump Inhibitor on the Single-Dose Pharmacokinetics of LOXO-292 in Healthy Adult Subjects

> Protocol No: LOXO-RET-18015 Final Protocol Date: 14 May 2018 Amendment 1 Date: 11 June 2018 Compound Name: LOXO-292

> > Celerion Project CA24336 Final Version 1.1 Date: 06 September 2018

Loxo Oncology, Inc. 701 Gateway Boulevard, Suite 420 South San Francisco, California 94080, USA

Celerion
621 Rose Street
Lincoln, Nebraska 68502, USA
And
100 Alexis-Nihon Boulevard, Suite 360,
Montreal, QC, H4M 2N8, Canada

Statistical Analysis Plan, Version 1.1, 06 September 2018


# Statistical Analysis Plan Signature Page

Compound Name: LOXO-292

Protocol: LOXO-RET-18015

Study Title: An Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food and a Proton Pump Inhibitor on the Single Dose Pharmacokinetics of LOXO-292 in Healthy Adult Subjects

Issue Date: 06 September 2018




# **Table of Contents**

| 1. | INT | RODUCTION | 6 |
|---|---|---|---|
| 2. | OBJ | ECTIVES AND ENDPOINTS | 6 |
| | 2.1 | Objectives | 6 |
| | 2.2 | Endpoints | 6 |
| 3. | STU | DY DESIGN | 7 |
| 4. | | ALYSIS POPULATIONS | |
| | 4.1 | Analysis Populations | |
| | 4.2 | Preliminary Data and Interim Analysis | |
| 5. | TRE | ATMENT DESCRIPTIONS | |
| 6. | | RMACOKINETIC ANALYSIS | |
| ٠. | 6.1 | Measurements and Collection Schedule | |
| | 6.2 | Bioanalytical Method for LOXO-292 | |
| | 6.3 | Investigational Product and PK Analyte Information of LOXO-292 | |
| | 6.4 | Pharmacokinetic Concentrations | |
| | 6.5 | Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292 | 11 |
| | 6.6 | Data Summarization and Presentation | |
| | 6.7 | Statistical Analysis of PK Parameters | |
| 7. | | ETY | |
| | 7.1 | Subject Discontinuation | |
| | 7.2 | Demographics | |
| | 7.3 | Adverse Events. | |
| | 7.4 | Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis) | |
| | 7.5 | Vital Signs (Blood Pressure, Pulse Rate, Respiration Rate, and Temperature) | |
| | 7.6 | ECG (Heart Rate, PR. ORS, OT, and OTcF [OT with Fridericia | |
| | | correction]) | |
| | 7.7 | Prior and Concomitant Medications | |
| | 7.8 | Physical Examination | |
| | 7.9 | Meals | |
| 8. | SUN | IMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 21 |
| 9. | SUN | IMARY TABLES AND FIGURES | |
| | 9.1 | In-text Summary Tables and Figures | |
| | 9.2 | Section 14 Summary Tables and Figures | |
| | 9.3 | Section 16 Data Listings | 26 |
| 10. | TAB | LE AND FIGURE SHELLS | 29 |

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18015 Celerion, Clinical Study Report No. CA24336

| 10.1 In-text Table Shells | 30 |
|-----------------------------|----|
| 10.2 Figures Shells | 35 |
| 10.3 Post-text Table Shells | |
| 11. LISTING SHELLS | 65 |

#### 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from study LOXO-RET-18015. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within the protocol or after the locking of the database will be documented in the clinical study report (CSR). The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data. Note that the header for this page will be the one used for the main body of the CSR.

Any additional exploratory analyses not addressed within this SAP and/or driven by the data, or requested by Loxo Oncology, Inc., will be considered out of scope and will be described in the CSR as needed.

#### 2. OBJECTIVES AND ENDPOINTS

#### 2.1 Objectives

# Primary:

- To assess the effect of food on the pharmacokinetics (PK) of LOXO-292 after a high fat meal in healthy adult subjects.
- To assess the effect of a gastric pH change on the PK of LOXO-292 after multiple doses of a proton pump inhibitor (PPI), omeprazole, under fasted and fed conditions in healthy adult subjects.

# Secondary:

To determine the safety and tolerability of a single dose of LOXO-292 with and without food, alone or in the presence of a PPI (omeprazole) in healthy adult subjects.

# 2.2 Endpoints

#### Pharmacokinetics:

The PK endpoints will include AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, CL/F, and t½ for LOXO-292 administered with and without food, and with and without PPI (omeprazole).

#### Safety:

Safety endpoints will include 12-lead electrocardiograms (ECGs), physical examinations, vital signs, clinical laboratory tests, and adverse events (AEs).


#### 3. STUDY DESIGN

This is an open label, randomized, 4-treatment, crossover study.

healthy, adult male and female subjects (women of non-childbearing potential only) were enrolled. Every attempt were made to enroll at least 3 subjects of each sex in the study.

Screening of subjects occurred within 28 days prior to the first dosing.

Subjects were randomized to one of four treatment sequences: ABCD, ABDC, BACD, and BADC. Every attempt was made to include the same number of females in each sequence and the same number of males in each sequence.

On Day 1 of Periods 1 and 2, a single oral dose of LOXO-292 was administered under fasted or fed conditions, according to the randomization schedule, followed by PK sampling for 168 hours.

In Periods 3 and 4, multiple oral doses of omeprazole were administered once daily from Day -4 of Period 3 until Day 7 of Period 4, inclusive (for a total of 18 consecutive days) with a single oral dose of LOXO-292 coadministered on Day 1 of each period under fasted or fed conditions, according to the randomization schedule. Pharmacokinetic sampling for LOXO-292 was taken for 168 hours following LOXO-292 dosing on Day 1 in each period.

There was a washout period of 7 days between LOXO-292 dose in Period 1 and LOXO-292 dose in Period 2 and between the LOXO-292 dose in Period 2 and the first dose of omeprazole in Period 3. There was no washout between Periods 3 and 4 omeprazole doses although the LOXO-292 doses will be separated by a 7-day washout.

Safety was monitored throughout the study by repeated clinical and laboratory evaluations.

Subjects were permitted to be replaced at the discretion of the Sponsor, but no subjects were replaced on this study.

Subjects were housed throughout the study beginning on Day -1 of Period 1, at the time indicated by the CRU, until after completion of the 168-hour blood draw and/or study procedures in Period 4. At all times, a subject may have been required to remain at the CRU for longer at the discretion of the Principal Investigator (PI) or designee.

The CRU made every attempt to contact all subjects who received at least 1 dose of study drug (including subjects who terminated the study early) using their standard procedures (i.e., phone call or other method of contact) approximately 7 days after the


last study drug administration (LOXO-292 or omeprazole, whichever came last) to determine if any AE had occurred since the last study visit.

# 4. ANALYSIS POPULATIONS

# 4.1 Analysis Populations

## **Safety Population**

All subjects who received at least one dose of LOXO-292 will be included in the safety evaluations.

# Pharmacokinetic Population

Samples from all subjects will be assayed even if the subjects do not complete the study. All subjects who comply sufficiently with the protocol and display an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations) will be included in the statistical analyses.

Data for each subject will be included in the summary statistics and statistical comparisons of PK parameters with the exceptions described as follows:

- Data from subjects who experience emesis at or before 2 times median Tmax for the given treatment during the PK sampling period time course of the study for LOXO-292 will be excluded from the summary statistics for the given treatment and from the statistical comparison of PK parameters.
- Data from subjects who significantly violate a protocol inclusion or exclusion criteria, deviate significantly from the protocol, or have unavailable or incomplete data which may influence the PK analysis will be excluded from the PK Population.

Any subject or data excluded from the analysis will be identified, along with their reason for exclusion, in the CSR.

## 4.2 Preliminary Data and Interim Analysis

No interim analysis is planned for this study.

#### 5. TREATMENT DESCRIPTIONS

LOXO-292 was supplied as 80 mg capsules.

Omeprazole was supplied as 40 mg delayed-release capsules.

All study drugs were administered orally with approximately 240 mL of water.

Subjects were instructed not to crush, split, or chew the study drugs.


Treatments A and B were dosed in Periods 1 and 2 and Treatments C and D were dosed in Periods 3 and 4 according to the randomization schedule. Treatments are described as follows:

# Periods 1 and 2:

# All Subjects CC

| Treatment | Short Description (text, tables headers, figures, listings, SAS output) | Abbreviated Description |
|---|---|---|
| A | 160 mg LOXO-292 fasted | 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions. |
| В | 160 mg LOXO-292 fed | 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast. |

# Periods 3 and 4:

Subjects were administered 40 mg of omeprazole (1 x 40 mg capsule) every 24 hours (within  $\pm$  1 hour of dosing time on Day -4 of Period 3) from Day -4 of Period 3 to Day 7 of Period 4, inclusive.

# All Subjects CCI

| Treatment | Short Description (text, tables headers, figures, listings, SAS output) | Abbreviated Description |
|---|---|---|
| С | Omeprazole + 160 mg LOXO-<br>292 fasted | Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions. |
| D | Omeprazole + 160 mg LOXO-<br>292 fed | Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat |

| breakfast. |
|------------|

For AEs, an additional treatment was added to account for the 4 days of omeprazole alone from Day -4 to Day -1 of Period 3.

| Treatment | Short Description (text, tables<br>headers, figures, listings, SAS<br>output) | Abbreviated Description |
|---|---|---|
| OMP<br>Alone | Omeprazole alone | Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3. |

#### 6. PHARMACOKINETIC ANALYSIS

#### 6.1 Measurements and Collection Schedule

Blood samples for PK assessment of LOXO-292 were taken at the following time points on Day 1 of each period: at predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose.

The 168-hour blood draw in Period 1 was the same as the predose blood draw in Period 2. The 168-hour blood draw in Period 3 was the same as the predose blood draw in Period 4.

All concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). However, if there were any significant deviations from nominal sample times, some concentration data may be excluded from mean concentration-time plots and/or additional concentration-time plots of the mean data may be provided. All deviations and excluded data will be provided and discussed in the CSR.

# 6.2 Bioanalytical Method for LOXO-292

Plasma concentrations of LOXO-292 were determined using a liquid chromatography-tandem mass spectrometry (LC-MS/MS) method validated with respect to accuracy, precision, linearity, sensitivity, and specificity at Alturas Analytics, Inc. (Moscow, Idaho, USA). The analytical range (lower limit of quantitation [LLOQ] – upper limit of quantitation [ULOQ]) for LOXO-292 is 1 – 1000 ng/mL. Samples that contain concentrations greater than 1000 ng/mL may have been diluted up to 51-fold, if necessary, to be within the quantification range.

# 6.3 Investigational Product and PK Analyte Information of LOXO-292

LOXO-292 has a molecular weight of approximately 500 g/mol. LOXO-292 was supplied as a powder-in-capsule containing 80 mg of drug substance (freebase) and as a simple blend with excipients in a hard gelatin capsule.

#### 6.4 Pharmacokinetic Concentrations

Plasma concentrations of LOXO-292 as determined at the collection times and per the bioanalytical method described in Section 6.1 and Section 6.2, respectively, will be used for the calculation of the plasma LOXO-292 PK parameters.

# 6.5 Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292

The appropriate noncompartmental PK parameters will be calculated from the plasma LOXO-292 concentration-time data using Phoenix WinNonlin Version 7.0 or higher. Actual sample times will be used in the calculations of the PK parameters. All PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Pharmacokinetic Parameters to be Calculated for LOXO-292

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| AUC0-t | Area under the concentration-time curve from time 0 to the time of the last observed non-zero concentration | Calculated using the<br>Linear Trapezoidal with<br>Linear Interpolation<br>Method |
| AUC0-inf | Area under the concentration-time curve from time 0 extrapolated to infinity | Calculated as AUC0-t + (Clast/Kel) where Clast is the last observed/measured concentration |
| AUC%extrap | Percent of AUC0-inf extrapolated | Calculated as<br>(1-AUC0-t/AUC0-<br>inf)*100 |
| Cmax | Maximum observed concentration | Taken directly from bioanalytical data |
| Tmax | The time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value | Taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax. |

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of<br>Determination |
|---|---|---|
| CL/F | Apparent total plasma clearance after oral (extravascular) administration | Calculated as<br>Dose/(AUC0-inf) |
| Kel | Apparent terminal elimination rate constant; represents the fraction of drug eliminated per unit time | Calculated as the negative of the slope of a linear regression of the log(concentration)-time for all concentrations > LLOQ |
| t½ | Apparent first-order terminal elimination half-life | Calculated as 0.693/Kel |

Pharmacokinetic parameters will not be calculated for subjects with fewer than 3 consecutive postdose time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from the statistical analysis.

For the calculation of the PK parameters, plasma concentrations below the limit of quantitation (BLQ) prior to the first quantifiable concentration will be set to 0 and plasma concentrations BLQ after the first quantifiable concentration will be treated as missing.

The Kel will be determined using linear regressions composed of at least 3 data points. The Kel will not be assigned if 1) the terminal elimination phase is not apparent, 2) if Tmax is one of the 3 last data points, or 3) if the R<sup>2</sup> value is less than 0.75. In cases where the Kel interval is not assigned, the values of t½, AUC0-inf, and CL/F are considered not calculable and will not be reported. Wherever the resulting t½ is more than half as long as the sampling interval, the Kel values and associated parameters (t½, AUC0-inf, AUC%extrap, and CL/F) may not be presented as judged appropriate and in accordance with Celerion SOPs.

If predose measurable concentrations were to occur, the following procedure will be used: if the predose concentration is less than or equal to 5% of Cmax for that subject period, the subject's data will be included in all PK measurements and calculations without any adjustments. If the predose value is greater than 5% of Cmax, the subject will be excluded from the PK analysis for that period only.

# 6.6 Data Summarization and Presentation

All LOXO-292 PK concentrations and PK parameters descriptive statistics will be generated using SAS<sup>®</sup> Version 9.3 or higher.

The plasma concentrations of LOXO-292 will be listed and summarized by treatment and time point for all subjects in the PK Population. Plasma concentrations of LOXO-


292 will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including sample size (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), standard error of the mean (SEM), minimum, median, and maximum will be calculated for all nominal concentration time points. Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

Mean and individual concentration-time profiles will be presented on linear and semilog scales. Linear mean plots will be presented with and without SD.

Plasma LOXO-292 PK parameters will be listed and summarized by treatment for all subjects in the PK Population. Pharmacokinetic parameters will be reported to 3 significant figures for individual parameters, with the exception of Tmax and t½, which will be presented with 2 decimal places. Summary statistics (n, Mean, SD, CV%, SEM, minimum, median, maximum, geometric mean [Geom Mean] and geometric CV% [Geom CV%]) will be calculated for plasma LOXO-292 PK parameters. Excluded subjects will be listed in the PK parameter tables, but will be excluded from the summary statistics and noted as such in the tables.

The level of precision for each concentration and PK parameter statistic will be presented as follows:

- minimum/maximum in same precision as in bioanalytical data and parameter output,
- mean/median in one more level of precision than minimum/maximum,
- SD/SEM in one more level of precision than mean/median,
- n will be presented as an integer, and
- CV% will be presented to the nearest tenth.

# 6.7 Statistical Analysis of PK Parameters

A comparison of In-transformed PK parameters (AUC0-t, AUC0-inf, and Cmax) will be made to evaluate the effect of:

- Food on the single-dose administration of LOXO-292 (Treatment B Versus Treatment A);
- The effect of gastric pH change by multiple-dose administrations of omeprazole on the single-dose administration of LOXO-292 under fasted conditions (Treatment C Versus Treatment A);


- The effect of gastric pH change by multiple-dose administrations of omeprazole on the single-dose administration of LOXO-292 under fed conditions (Treatment D Versus Treatment B);
- The effect of food on the single-dose administration of LOXO-292 under gastric pH change by multiple-dose administrations of omeprazole (Treatment D Versus Treatment C)

by performing an analysis of variance (ANOVA) model using PROC MIXED in  $SAS^{@}$ .





#### 7. SAFETY

No inferential statistics are to be performed for the safety analysis.

All clinical safety and tolerability data will be listed by subject and assessment time points, including rechecks, unscheduled assessments, and early termination (ET), chronologically.

Continuous variables will be summarized using n, arithmetic mean, SD, minimum, median, and maximum. Frequency counts will be reported for categorical data when appropriate.


The level of precision will be presented as follows: "n" as an integer, minimum/maximum in same precision as in the database, mean/median in one more precision level than minimum/maximum, and SD in one more precision level than mean/median.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

When change from baseline is calculated, baseline is the last scheduled assessment before dosing of LOXO-292 at each period, including rechecks and unscheduled assessments, whichever is later, unless otherwise specified in the sections below. Rechecks, unscheduled assessments and ET measurements taken after first dosing will not be used in the summarization.

## 7.1 Subject Discontinuation

Subjects will be summarized by the number of subjects enrolled, completed, and discontinued from the study with discontinuation reasons by treatment sequence and overall. Individual subject's dosing status for each treatment will be provided along with their study completion status and date. Disposition data will be listed by subject.

# 7.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index) by treatment sequence and overall. Weight, height and body mass index are summarized at screening. Age will be derived from the date of birth to the date of first dosing. Frequency counts will be provided for categorical variables (race, ethnicity, and sex). A by-subject listing will also be provided.

#### 7.3 Adverse Events

All adverse events (AEs) occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 21.0.

Each AE will be graded, by the clinical site, on the National Institution of Health's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) 5-point severity scale (Grades 1, 2, 3, 4 and 5). Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection. The following definitions for clinical descriptions of severity grade for each AE are based on the following general guideline [CTCAE Nov 2017]:

Table 7.3: Adverse Event Severity Grade Level and Description

| Grade | Description |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL*. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE. |

<sup>\*</sup> Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

Similarly, the causal relationship of the study drugs to the AE will be described as Related or Unrelated to study drugs LOXO-292 and/or omeprazole.

All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, treatment group, severity grade, relationship to study drugs, and action; however, only treatment-emergent AEs (TEAEs) will be summarized.

A TEAE is defined as an undesirable event not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. Each TEAE will be attributed to a treatment based on investigator judgment as well as its onset date and time. An AE that occurs during the washout period between treatments will be considered treatment-emergent to the last treatment given. If an AE has a change in severity grade, the original AE will be given a resolution date and time, of the time of severity grade increase or decrease, and a new AE record will be initiated with the new severity grade, and the new AE record will use the resolved date/time of the previous record as onset date/time. If an AE decreases in severity grade, the new AE record with less severity will be considered and counted as the same AE event of the previous record with worse severity under

<sup>\*\*</sup> Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications and not bedridden.

the same treatment group and period in the analysis and summary tables. If the severity of an AE remains the same, the AE will be kept open through to resolution.

If the onset time of an AE is missing and the onset date is the same as the LOXO-292 treatment dosing date, then the AE will be considered treatment-emergent in both the prior and current treatment. If the onset time of an AE is missing and the onset date does not fall on a LOXO-292 dosing date, then the AE will be considered treatment-emergent for the last treatment administered. If the onset date of an AE is missing, then the AE will be considered treatment-emergent and attributed to the first treatment group on the study, unless the onset date is known to have occurred within or between specific treatment periods.

TEAEs will be tabulated by system organ class and preferred term. Summary tables will include the number of subjects reporting the AE and as a percent of the number of subjects dosed by treatment and overall. In addition to the protocol defined Treatments A, B, C, D, an additional treatment OMP Alone will be used to account for the time period of omeprazole administered alone, i.e., multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3. In addition, the number of AEs will be summarized. Tables will also be presented by severity grade and relationship to study drugs. If a subject experienced the same TEAE more than once with different level of severity grade for a given treatment, only the most severe one will be counted. Similarly, if a subject experienced the same TEAE more than once with different level of drug relationship for a given treatment, only the one most closely related to the study drug will be counted.

Should any serious adverse events (SAEs) occur during the study, the SAEs will be displayed in a table and a narrative included in the Clinical Study Report.

# 7.4 Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis)

All clinical laboratory test results will be presented in by-subject data listings, however, only serum chemistry, hematology, coagulation and urinalysis values will be summarized.

Hematology, coagulation, serum chemistry and urinalysis tests will be conducted at the following time points:

**Table 7.4 Lab Test Time Points** 

| Period | Period Day |
|--------|------------|
| Screen | Screening |
| 1 | Day -1* |
| 1 | Day 4* |
| 1 | Day 7* |

| 2 | Day 4* |
|---|---|
| 2 | Day 7* |
| 3 | Day 4** |
| 3 | Day 7** |
| 4 | Day 4** |
| 4 | Day 8*** |
| * performe | ed following a fast of at least 8 hours |
| ** performed prior dosing of omeprazole | |
| *** performed at the end of Period 4 or prior to | |

Early Termination (ET)

Out-of-normal range (OOR) flags will be recorded as follows: high (H) and low (L) for numerical results and did-not-match (\*) for categorical results. If a value fails the reference range, it will automatically be compared to a computer clinically significant (CS) range suggested by the PI (Celerion SOP GSOP.10.1028). If the value falls within the computer CS range, it will be noted as "N" for not clinically significant. If the value fails (i.e. falls outside of the CS range) the computer CS range, it will be flagged with a "Y" which prompts the PI to determine how the OOR value should be followed using 4 Investigator flags: "N", not clinically significant, "R", requesting a recheck, "^", checking at the next scheduled visit, or "Y", clinically significant. To distinguish the PI flag from the CS range flags, the PI flags "N" and "Y" will be presented as "-" and "+" in the data listings, respectively. Additionally, a derived flag based on a search of the PI comments for a comment of "CS" or "Clinically Significant" will be used. The derived flag will be populated with "+" if the positive clinically significant determination is found in the comments for cases when the PI flag is populated with a "^" or an "R". In addition, CTCAE Version 5.0 grading (found in NCI CTCAE guidance) will be applied to all out-of-range lab values deemed clinically significant by the investigator or designee which are recorded as AEs. The resulting flag, e.g., G1, will be placed along with the Celerion flags (see shell of Table 14.3.4.4).

Out-of-range values and corresponding recheck results will be listed. Other lab results within this panel and time point will also be listed for this subject. Results that are indicated as CS by the PI (either in the PI flag or in PI comments) will be listed in the table. Out-of-range values laboratory value results which are indicated as CS by the PI will be reported as AEs.

For all laboratory values that are numeric, descriptive statistics (n, mean, SD, minimum, median, and maximum) will be presented for each laboratory test by treatment and time point. Change from baseline (defined below) will also be summarized. In general, postdose unscheduled events or rechecks will not be summarized. Similarly, ET results will not be included in summaries.

For each laboratory test, a shift table will be developed comparing the frequency of the results at baseline (above normal, normal, or below normal) to postdose results for


each part, respectively. For urinalysis tests, the categories are normal and outside normal.

Baseline is Day -1 of Period 1 and Day 7 of previous period for Period 2, 3, 4 and is the last non-missing predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments. Day 7 measurement of Period 1, 2, 3 might be used twice as postdose value of Period 1, 2, 3 and baseline value of Period 2, 3, 4. When serving as baseline of Period 2, 3, 4, the re-check or unscheduled values after Day 7 of Period 1, 2, 3 and prior to LOXO-292 dosing of Period 2, 3, 4 could be used as baseline.

#### 7.5 Vital Signs (Blood Pressure, Pulse Rate, Respiration Rate, and Temperature)

Vital signs were performed at the following time points:

**Table 7.5 Vital Signs Time Points** 

| ameter |
|-----------|
| BP, RR, T |
| , BP, RR |
| BP, RR, T |
| , |

Descriptive statistics will be reported for vital sign measurements (blood pressure, pulse, and respiration rate) and change from baseline by treatment and time point. Baseline is Day -1 of Period 1 and Day 1 predose of Period 2, 3, 4 and is the last nonmissing predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments. Postdose recheck values and ET results will not be used for calculation of descriptive statistics. All vital signs results will be listed by subject.

<sup>\*\*</sup> performed prior dosing

<sup>\*\*\*</sup> performed at the end of Period 4 or prior to ET

#### 7.6 ECG (Heart Rate, PR, QRS, QT, and QTcF [QT with Fridericia correction])

Single 12-lead ECGs were performed at the following time points:

**Table 7.6: ECG Time Points** 

| Period | Period Day | Study Hour |
|------------------------------------------|------------|------------|
| Screen | Screening | |
| 1 | Day -1 | 0* |
| 1 | Day 1 | 2 |
| 1 | Day 4 | 72 |
| 2 | Day 1 | 0** |
| 2 | Day 1 | 2 |
| 2 | Day 4 | 72 |
| 3 | Day 1 | 0** |
| 3 | Day 1 | 2 |
| 3 | Day 4 | 72 |
| 4 | Day 1 | 0** |
| 4 | Day 1 | 2 |
| 4 | Day 4 | 72 |
| 4 | Day 8 | 168*** |
| * performed within 24 hours prior dosing | | |

<sup>\*\*</sup> performed prior dosing

Descriptive statistics will be reported for ECG parameters and change from baseline by treatment and time point. Baseline is Day -1 of Period 1 and Day 1 predose of Period 2, 3, 4 and is the last non-missing predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments. Postdose recheck values and ET results will not be used for calculation of descriptive statistics. QTcF values that are > 450 msec and increase from baseline > 30 msec will be flagged in the data listing. All ECG interval parameters will be listed by subject and time point of collection.

# 7.7 Prior and Concomitant Medications

All prior concomitant medications recorded during the study will be coded with the WHO Dictionary, Version Mar2017 B3 and listed. Note: Per Exclusion Criterion 15, subjects should refrain from using any drug, including prescription and non-prescription medications, herbal remedies, and vitamin supplements 14 days prior to the first dosing and throughout the study. After dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee.

<sup>\*\*\*</sup> performed at the end of Period 4 or prior to ET

#### 7.8 Physical Examination

Physical examinations will be performed at screening. Abbreviated physical examinations may be performed at check-in (Day -1) of the first period. Abnormal findings will be reported as medical history or adverse events by the clinical site. Physical examination results will be listed by subject and time point.

#### 7.9 Meals

The composition of meals will be provided in the CSR. If the subject only eats part of the meal, the percentage of meals that is not consumed will be documented in the comment field of the Meal Times dataset.

#### 8. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol.

#### 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Council for Harmonisation (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using SAS<sup>®</sup> Version 9.3 or higher.

# 9.1 In-text Summary Tables and Figures

The following is a list of table and figure titles that will be included in the text of the CSR. Tables and figures will be numbered appropriately during compilation of the CSR.

#### Section 10:

Table 10-1 Summary of Disposition (Safety Population)

# Section 11:

Table 11-1 Demographic Summary (Safety Population)

# Table 11-2 Summary of Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of 160 mg LOXO-292 Fasted (Treatment A), Administration of 160 mg LOXO-292 Fed (Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C), and Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) (Pharmacokinetic Population)

- Table 11-3 Summary of Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of 160 mg
  LOXO-292 Fed (Treatment B) Versus Administration of 160 mg
  LOXO-292 Fasted (Treatment A) (Pharmacokinetic Population)
- Table 11-4 Summary of Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Coadministration of Multiple
  Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C) Versus
  Administration of 160 mg LOXO-292 Fasted (Treatment A)
  (Pharmacokinetic Population)
- Table 11-5 Summary of Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Coadministration of Multiple
  Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) Versus
  Administration of 160 mg LOXO-292 Fed (Treatment B)
  (Pharmacokinetic Population)
- Table 11-6 Summary of Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Coadministration of Multiple
  Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) Versus
  Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292
  Fasted (Treatment C) (Pharmacokinetic Population)
- Figure 11-1 Arithmetic Mean Plasma LOXO-292 Concentration-Time Profiles
  Following Administration of 160 mg LOXO-292 Fasted (Treatment
  A), Administration of 160 mg LOXO-292 Fed (Treatment B),
  Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292
  Fasted (Treatment C), and Coadministration of Multiple Dose
  Omeprazole + 160 mg LOXO-292 Fed (Treatment D)
  (Pharmacokinetic Population)

# Section 12:

Table 12-1 Treatment-Emergent Adverse Event Frequency by Treatment – Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

# 9.2 Section 14 Summary Tables and Figures

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be renumbered as appropriate during the compilation of the report.

# 14.1 Demographic Data Summary Tables

#### 14.1.1 Demographic Tables

| Table 14.1.1.1 | Summary of Disposition (Safety Population) |
|----------------|---------------------------------------------|
| Table 14.1.1.2 | Disposition of Subjects (Safety Population) |
| Table 14.1.1.3 | Demographic Summary (Safety Population) |

# 14.2 Pharmacokinetic Data Summary Tables and Figures

| | v e |
|---|---|
| 14.2.1 Plas | ma LOXO-292 Tables |
| Table 14.2.1.1 | Plasma LOXO-292 Concentrations (ng/mL) Following<br>Administration of 160 mg LOXO-292 Fasted (Treatment<br>A) (Pharmacokinetic Population) |
| Table 14.2.1.2 | Plasma LOXO-292 Concentrations (ng/mL) Following<br>Administration of 160 mg LOXO-292 Fed (Treatment B)<br>(Pharmacokinetic Population) |
| Table 14.2.1.3 | Plasma LOXO-292 Concentrations (ng/mL) Following<br>Coadministration of Multiple Dose Omeprazole + 160 mg<br>LOXO-292 Fasted (Treatment C) (Pharmacokinetic<br>Population) |
| Table 14.2.1.4 | Plasma LOXO-292 Concentrations (ng/mL) Following<br>Coadministration of Multiple Dose Omeprazole + 160 mg<br>LOXO-292 Fed (Treatment D) (Pharmacokinetic<br>Population) |
| Table 14.2.1.5 | Plasma LOXO-292 Pharmacokinetic Parameters Following<br>Administration of 160 mg LOXO-292 Fasted (Treatment<br>A) (Pharmacokinetic Population) |
| Table 14.2.1.6 | Plasma LOXO-292 Pharmacokinetic Parameters Following<br>Administration of 160 mg LOXO-292 Fed (Treatment B)<br>(Pharmacokinetic Population) |
| Table 14.2.1.7 | Plasma LOXO-292 Pharmacokinetic Parameters Following<br>Coadministration of Multiple Dose Omeprazole + 160 mg<br>LOXO-292 Fasted (Treatment C) (Pharmacokinetic<br>Population) |

| Table 14.2.1.8 | Plasma LOXO-292 Pharmacokinetic Parameters Following |
|----------------|-------------------------------------------------------|
| | Coadministration of Multiple Dose Omeprazole + 160 mg |
| | LOXO-292 Fed (Treatment D) (Pharmacokinetic |
| | Population) |

Table 14.2.1.9 Intervals (Hours) Used for Determination of Plasma
LOXO-292 Kel Values Following Administration of 160
mg LOXO-292 Fasted (Treatment A), Administration of
160 mg LOXO-292 Fed (Treatment B), Coadministration
of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted
(Treatment C), and Coadministration of Multiple Dose
Omeprazole + 160 mg LOXO-292 Fed (Treatment D)
(Pharmacokinetic Population)

- Table 14.2.1.10 Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Administration of
  160 mg LOXO-292 Fed (Treatment B) Versus
  Administration of 160 mg LOXO-292 Fasted (Treatment
  A) (Pharmacokinetic Population)
- Table 14.2.1.11 Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Coadministration
  of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted
  (Treatment C) Versus Administration of 160 mg LOXO292 Fasted (Treatment A) (Pharmacokinetic Population)
- Table 14.2.1.12 Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Coadministration
  of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed
  (Treatment D) Versus Administration of 160 mg LOXO292 Fed (Treatment B) (Pharmacokinetic Population)
- Table 14.2.1.13 Statistical Comparisons of Plasma LOXO-292
  Pharmacokinetic Parameters Following Coadministration
  of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed
  (Treatment D) Versus Coadministration of Multiple Dose
  Omeprazole + 160 mg LOXO-292 Fasted (Treatment C)
  (Pharmacokinetic Population)

# 14.2.2 Plasma LOXO-292 Figures

- Figure 14.2.2.1 Mean (SD) Plasma LOXO-292 Concentration-Time
  Profiles Following Administration of 160 mg LOXO-292
  Fasted (Treatment A), Administration of 160 mg LOXO292 Fed (Treatment B), Coadministration of Multiple Dose
  Omeprazole + 160 mg LOXO-292 Fasted (Treatment C),
  and Coadministration of Multiple Dose Omeprazole + 160
  mg LOXO-292 Fed (Treatment D) (Linear Scale)
  (Pharmacokinetic Population)
- Figure 14.2.2.2 Mean Plasma LOXO-292 Concentration-Time Profiles
  Following Administration of 160 mg LOXO-292 Fasted
  (Treatment A), Administration of 160 mg LOXO-292 Fed
  (Treatment B), Coadministration of Multiple Dose
  Omeprazole + 160 mg LOXO-292 Fasted (Treatment C),
  and Coadministration of Multiple Dose Omeprazole + 160
  mg LOXO-292 Fed (Treatment D) (Linear Scale)
  (Pharmacokinetic Population)
- Figure 14.2.2.3 Mean Plasma LOXO-292 Concentration-Time Profiles
  Following Administration of 160 mg LOXO-292 Fasted
  (Treatment A), Administration of 160 mg LOXO-292 Fed

(Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C), and Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) (Semi-Log Scale) (Pharmacokinetic Population)

# 14.3 Safety Data Summary Tables

# 14.3.1 Displays of Adverse Events

- Table 14.3.1.1 Treatment-emergent Adverse Event Frequency by Treatment
   Number of Subjects Reporting Events (% of Subject
  Dosed) (Safety Population)
- Table 14.3.1.2 Treatment-emergent Adverse Event Frequency by Treatment
   Number of Adverse Events (% of Total Adverse Events)
  (Safety Population)
- Table 14.3.1.3 Treatment-Emergent Adverse Event Frequency by
  Treatment, Severity Grade, and Relationship to Study Drugs
   Number of Subjects Reporting Events (Safety Population)
- Table 14.3.1.4 Treatment-Emergent Adverse Event Frequency by
  Treatment, Severity Grade, and Relationship to Study Drugs
   Number of Adverse Events (Safety Population)

#### 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population)
<if no serious adverse event occurred, a statement 'There was no serious adverse event recorded during the study." will be added>

# 14.3.3. Narratives of Deaths, other Serious and Certain other Significant Adverse Events

# 14.3.4. Abnormal Laboratory Value Listing (each patient)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry (Safety Population)
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology and Coagulation
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Urinalysis
- Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

# 14.3.5. Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline –
Serum Chemistry (Safety Population)

Table 14.3.5.2 Clinical Laboratory Shift from Baseline – Serum Chemistry (Safety Population)

Table 14.3.5.3 Clinical Laboratory Summary and Change from Baseline –
Hematology and Coagulation (Safety Population)

Table 14.3.5.4 Clinical Laboratory Shift from Baseline – Hematology and Coagulation (Safety Population)

Table 14.3.5.5 Clinical Laboratory Summary and Change from Baseline –
Urinalysis (Safety Population)

Table 14.3.5.6 Clinical Laboratory Shift from Baseline – Urinalysis (Safety Population)

Table 14.3.5.7 Vital Sign Summary and Change from Baseline (Safety Population)

Table 14.3.5.8 12-Lead Electrocardiogram Summary and Change from

# 9.3 Section 16 Data Listings

Note: Virology test results (Hepatitis and HIV) that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in the database transfer.

Baseline (Safety Population)

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

#### 16.1 Study Information

Appendix 16.1.9 Statistical Methods

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

# 16.2. Subject Data Listings

#### 16.2.1. Subject Discontinuation

Appendix 16.2.1 Subject Discontinuation (Safety Population)

#### 16.2.2. Protocol Deviations

Appendix 16.2.2 Protocol Deviations

# 16.2.3. Subjects Excluded from Pharmacokinetic Analysis

Appendix 16.2.3 Subjects Excluded from Pharmacokinetic Analysis

Note: Appendices 16.2.2 and 16.2.3 are generated in MS Word for inclusion in the CSR.

# 16.2.4 Demographic Data

| Appendix 16.2.4.1 | Demographics (Safety Population) |
|-------------------|--------------------------------------------------|
| Appendix 16.2.4.2 | Updated Informed Consent (Safety Population) |
| Appendix 16.2.4.3 | Physical Examination (Safety Population) |
| Appendix 16.2.4.4 | Medical and Surgical History (Safety Population) |
| Appendix 16.2.4.5 | Nicotine Use (Safety Population) |

# 16.2.5. Compliance and Drug Concentration Data

| 10.2.5. Comphane | e and Drug Concentration Data |
|---------------------|--------------------------------------------------------|
| Appendix 16.2.5.1.1 | Inclusion Criteria |
| Appendix 16.2.5.1.2 | Exclusion Criteria |
| Appendix 16.2.5.2 | Subject Eligibility (Safety Population) |
| Appendix 16.2.5.3.1 | Check-in and Return Criteria |
| Appendix 16.2.5.3.2 | Check-in and Return Responses (Safety Population) |
| Appendix 16.2.5.4.1 | Test Compound Description |
| Appendix 16.2.5.4.2 | Test Compound Administration Times (Safety Population) |
| Appendix 16.2.5.5 | PK Blood Draw Times (Safety Population) |
| Appendix 16.2.5.6 | Phone Call (Safety Population) |
| Appendix 16.2.5.7 | Meal Times (Safety Population) |
| Appendix 16.2.5.8 | Prior and Concomitant Medications (Safety Population) |

# 16.2.6 Individual Pharmacokinetic Response Data

| Appendix 16.2.6 | Individual Plasma LOXO-292 Concentration Versus |
|-----------------|----------------------------------------------------|
| | Time Profiles Following Administration of 160 mg |
| | LOXO-292 Fasted (Treatment A), Administration of |
| | 160 mg LOXO-292 Fed (Treatment B), |
| | Coadministration of Multiple Dose Omeprazole + 160 |
| | mg LOXO-292 Fasted (Treatment C), and |
| | Coadministration of Multiple Dose Omeprazole + 160 |
| | mg LOXO-292 Fed (Treatment D) for Subject X |
| | (Linear and Semi-Log Scale) |

# 16.2.7 Adverse Events Listings

| Appendix 16.2.7.1 | Adverse Events (I of II) (Safety Population) |
|---|---|
| Appendix 16.2.7.2 | Adverse Events (II of II) (Safety Population) |
| Appendix 16.2.7.3 | Adverse Event Non-Drug Therapy (Safety Population) |
| Appendix 16.2.7.4 | Adverse Event Preferred Term Classification (Safety Population) |

# 16.2.8 Listings of Individual Laboratory Measurements and Other Safety Observations

| Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry (Safety Population) |
|---|---|
| Appendix 16.2.8.1.2 | Clinical Laboratory Report - Hematology and<br>Coagulation (Safety Population) |
| Appendix 16.2.8.1.3 | Clinical Laboratory Report - Urinalysis (Safety Population) |
| Appendix 16.2.8.1.4 | Clinical Laboratory Report - Urine Drug Screening (Safety Population) |
| Appendix 16.2.8.1.5 | Clinical Laboratory Report - Comments (Safety Population) |
| Appendix 16.2.8.2 | Vital Signs (Safety Population) |
| Appendix 16.2.8.3 | 12-Lead Electrocardiogram (Safety Population) |

#### 10. TABLE AND FIGURE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables and figures that will be presented and included in the final CSR. Unless otherwise noted, all in-text tables will be presented in Times New Roman font size 8 and post-text tables in Courier New font size 9. These tables will be generated according to the ADaM Model 2.1 and ADaM implementation guide 1.1.

#### 10.1 In-text Table Shells

# Table 10-1 Summary of Disposition (Safety Population)

| Disposition | ABCD | ABDC | BACD | BADC | Overall |
|---|---|---|---|---|---|
| Enrolled | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Completed Study | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Discontinued Early | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| <reason1></reason1> | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| <reason2></reason2> | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions. Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Source: Table 14.1.1.1

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_disp.sas DDMMMYYYY HH:MM

Table 11-1 Demographic Summary (Safety Population)

| | | Treatment Sequence | | | | |
|---|---|---|---|---|---|---|
| Trait | | ABCD | ABDC | BACD | BADC | Overall |
| Sex | Male | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Female | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Race | Asian | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Black or African American | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | White | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Ethnicity | Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Not Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Age* (yr) | n | XX | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Height (cm) | n | XX | XX | XX | XX | XX |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XXX | XXX | XXX | XXX | XXX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Maximum | XXX | XXX | XXX | XXX | XXX |

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

\* Age is calculated from the date of first dosing.

BMI = Body mass index

Source: Table 14.1.1.3

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_dem.sas DDMMMYYYY HH:MM

**Programmer Note:** Weight (kg) and BMI (kg/m<sup>2</sup>) will also be summarized in the table above.

In-text Table 11-2 will be in the following format:

Table 11-2 Summary of Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of 160 mg LOXO-292 Fasted (Treatment A), Administration of 160 mg LOXO-292 Fed (Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) (Pharmacokinetic Population)

| Pharmacokinetic Parameters | Treatment A | Treatment B | Treatment C | Treatment D |
|---|---|---|---|---|
| Param1 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param2 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param3 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param4 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

AUCs and Cmax values are presented as geometric mean (geometric CV%).

Tmax values are presented as median (min, max).

Other parameters are presented as arithmetic mean  $\pm$  SD.

Source: Tables 14.2.1.5 through 14.2.1.8

# Notes for Generating the Actual Table:

Presentation of Data:

- The following PK parameters will be presented in the following order: AUC0-t <unit>, AUC0-inf <unit>, AUC%extrap <unit>, Cmax <unit>, Tmax <unit>, Kel <unit>, and CL/F <unit>
- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells

Program: /CAXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM


In-text Tables 11-3 through 11-6 will be in the following format:

Table 11-3 Summary of Statistical Comparisons of Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of 160 mg LOXO-292 Fed (Treatment B) Versus Administration of 160 mg LOXO-292 Fasted (Treatment A) (Pharmacokinetic Population)

| | Treatment B (Test) | | Treatment A (Reference) | | GMR (%) | 90% Confidence<br>Interval | Intra-subject<br>CV% |
|---|---|---|---|---|---|---|---|
| Parameter | Geometric LSMs | n | Geometric LSMs | n | | | |
| param1 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX | X.XX |
| param2 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX | X.XX |
| param3 (units) | XXX.X | XX | XXX.X | XX | XX.XX | XX.XX - XX.XX | X.XX |

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Geometric least-squares means (LSMs) are calculated by exponentiating the LSMs derived from the ANOVA.

Geometric Mean Ratio (GMR) = 100\*(test/reference)

Intra-subject CV% was calculated as 100 x square root(exp[MSE]-1), where MSE = Residual variance from ANOVA.

Source: Table 14.2.1.10

#### **Notes for Generating the Actual Table:**

#### Presentation of Data:

- The following PK parameters will be presented in the following order: AUC0-t
   <unit>, AUC0-inf <unit>, and Cmax <unit>
- n will be presented as an integer (with no decimal);
- All statistics will be presented with same precision as defined in post-text shells

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM

Table 12-1 Treatment-Emergent Adverse Event Frequency by Treatment – Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

| Adverse Events* | A | В | OMP Alone<br>XX (100%) | C<br>XX (100%) | <b>D</b> XX (100%) | Overall<br>XX (100%) |
|---|---|---|---|---|---|---|
| Number of Subjects Dosed | XX (100%) | XX (100%) | | | | |
| Number of Subjects With TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects Without TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| System Organ Class 1 | X (X%) | X (X%) | X ( X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 1 | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 2 | X (X%) | X (X%) | X ( X%) | X (X%) | X (X%) | X (X%) |
| System Organ Class 2 | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 1 | X (X%) | X (X%) | X ( X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 2 | X (X%) | X (X%) | X ( X%) | X (X%) | X (X%) | X (X%) |

\*Adverse events are coded using MedDRA® Version 21.0 by System Organ Class and Preferred Term.

TEAE = Treatment-emergent Adverse event

Although a subject may have had 2 or more clinical adverse experiences, the subject is counted only once within a category. The same subject may appear in different categories.

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat

Treatment OMP Alone: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80

mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

Source: Table 14.3.1.1

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_ae.sas DDMMMYYYY HH:MM

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column.

# 10.2 Figures Shells

In-text Figure 11-1 and Figure 14.2.2.2 will be in the following format:

Figure 11-1 Arithmetic Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of 160 mg LOXO-292 Fasted (Treatment A), Administration of 160 mg LOXO-292 Fed (Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C), and Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) (Pharmacokinetic Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

Statistical Analysis Plan, 06 September 2018


### Notes for Generating the Actual Mean Figure:

- Legend will be:
  - o Treatment A: 160 mg LOXO-292 fasted
  - o Treatment B: 160 mg LOXO-292 fed
  - o Treatment C: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fasted
  - o Treatment D: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fed
- Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)" for all figures
- X-axis label will be "Hours post LOXO-292 dose (hr)" for all figures
- Add footnote: LLOQ value for LOXO-292 is 1 ng/mL

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMYYYY HH:MM

Figure 14.2.2.1 will be in the following format:

Figure 14.2.2.1 Mean (SD) Plasma LOXO-292 Concentration-Time Profiles Following Administration of 160 mg LOXO-292 Fasted (Treatment A), Administration of 160 mg LOXO-292 Fed (Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C), and Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) (Linear Scale) (Pharmacokinetic Population)



Statistical Analysis Plan, 06 September 2018


### Notes for Generating the Actual Mean Figure:

- Legend will be:
  - o Treatment A: 160 mg LOXO-292 fasted
  - o Treatment B: 160 mg LOXO-292 fed
  - o Treatment C: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fasted
  - o Treatment D: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fed
- Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)" for all figures
- X-axis label will be "Hours post LOXO-292 dose (hr)" for all figures
- Add footnote: LLOQ value for LOXO-292 is 1 ng/mL

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMYYYY HH:MM

Figure 14.2.2.3 will be in the following format:

Figure 14.2.2.3 Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of 160 mg LOXO-292 Fasted (Treatment A), Administration of 160 mg LOXO-292 Fed (Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C), and Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) (Semi-Log Scale) (Pharmacokinetic Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

Statistical Analysis Plan, 06 September 2018


### Notes for Generating the Actual Mean Figure:

- Legend will be:
  - o Treatment A: 160 mg LOXO-292 fasted
  - o Treatment B: 160 mg LOXO-292 fed
  - o Treatment C: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fasted
  - o Treatment D: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fed
- Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)" for all figures
- X-axis label will be "Hours post LOXO-292 dose (hr)" for all figures
- Add footnote: LLOQ value for LOXO-292 is 1 ng/mL

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMYYYY HH:MM

Appendix 16.2.6 will be in the following format:

## Appendix 16.2.6

Individual Plasma LOXO-292 Concentration Versus Time Profiles Following Administration of 160 mg LOXO-292 Fasted (Treatment A), Administration of 160 mg LOXO-292 Fed (Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C), and Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) for Subject X (Linear and Semi-Log Scale)



Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMMYYY HH:MM

Statistical Analysis Plan, 06 September 2018


#### Notes for Generating the Actual Mean Figure:

- Legend will be:
  - o Treatment A: 160 mg LOXO-292 fasted
  - o Treatment B: 160 mg LOXO-292 fed
  - Treatment C: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fasted
  - o Treatment D: 40 mg multiple daily doses of omeprazole + 160 mg LOXO-292 fed
- Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)" for all figures
- X-axis label will be "Hours post LOXO-292 dose (hr)" for all figures
- Add footnote: LLOQ value for LOXO-292 is 1 ng/mL

Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMYYYYY HH:MM

#### 10.3 Post-text Table Shells

Page X of X

Table 14.1.1.1 Summary of Disposition (Safety Population)

| Disposition | ABCD | ABDC | BACD | BADC | Overall |
|---|---|---|---|---|---|
| Enrolled<br>Completed<br>Discontinued Early<br>Reason 1<br>Reason 2<br>Reason 3<br>etc. | XX<br>XX<br>XX<br>XX<br>XX | XX<br>XX<br>XX<br>XX<br>XX<br>XX | XX<br>XX<br>XX<br>XX<br>XX<br>XX | XX<br>XX<br>XX<br>XX<br>XX | XX<br>XX<br>XX<br>XX<br>XX |

Note: Treatment A: 160 mg LCXC-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg comprazole (1  $\times$  40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2  $\times$  80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Page X of X

Table 14.1.1.2 Disposition of Subjects (Safety Population)

| | | | | ment Dos | | | | | ent Comp | | | Study Completion | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Randomized<br>Sequence | A | В | OMP<br>Alone | | D | A | В | OMP<br>Alone | | D | Status | Date |
| XXX-XXX<br>XXX-XXX | ABCD<br>ABDC | Yes<br>Yes | Yes<br>Yes | Yes<br>No | Yes<br>No | Yes<br>No | Yes<br>Yes | Yes<br>Yes | Yes<br>No | Yes<br>No | Yes<br>No | Completed Study Terminated Study Prematurely | DDMMYYYY<br>DDMMYYYY |

Note: Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment OMP Alone: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg

capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM


Table 14.1.1.3 Demographic Summary (Safety Population)

| Trait | | ABCD | ABDC | BACD | BADC | Overall |
|---|---|---|---|---|---|---|
| Sex | Male<br>Female | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) | X ( XX%) |
| Race | Asian<br>Black or African American<br>White | X ( XX%)<br>X ( XX%) | | X ( XX%)<br>X ( XX%)<br>X ( XX%) | X ( XX%)<br>X ( XX%)<br>X ( XX%) | X ( XX%)<br>X ( XX%)<br>X ( XX%) |
| Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | X ( XX%) | X ( XX%)<br>X ( XX%) | X ( XX%)<br>X ( XX%) | X ( XX%) | X ( XX%) |
| Age*(yr) | n<br>Mean<br>SD<br>Median<br>Minimum<br>Maximum | XX<br>XX.X<br>X.XX<br>XX.X<br>XX<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX<br>XX | XX<br>XX.X<br>X.XX<br>XX.X<br>XX<br>XX |
| Height (cm) | n<br>Mean<br>SD<br>Median<br>Minimum<br>Maximum | XX<br>XX.XX<br>XX.XXX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.XX<br>XX.XXX<br>XX.X<br>XX.X<br>XX.X | XX<br>XX.XX<br>XX.XX<br>XX.X<br>XX.X | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.X<br>XX.X | XX<br>XX.XX<br>XX.XXX<br>XX.XX<br>XX.X<br>XX.X |

**Programmer Note:** Also include weight (kg) and BMI (kg/m²)

Note: \* Age is calculated from the date of first dosing. BMI = Body mass index

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment C: Multiple daily doses of 40 mg omeprazole (1  $\times$  40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2  $\times$  80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg comeprazole (1  $\times$  40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2  $\times$  80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


## Tables 14.2.1.1 through 14.2.1.4 will be in the following format:

Table 14.2.1.1 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of 160 mg LOXO-292 Fasted (Treatment A) (Pharmacokinetic Population)

| | | | (hr) | le Times | Samp | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Study | Treatment | Subject |
| XX | XX | XX | XX | XX | XX | XX | XX | Predose | Period | Sequence | Number |
| XX | XX | XX | XX | XX | XX | XX | XX | BLQ | Х | XXX | XXX-XXX |
| XX | XX | XX | XX | XX | XX | XX | XX | BLQ | X | XXX | XXX-XXX |
| XX | XX | XX | XX | XX | XX | XX | XX | BLQ | X | XXX | XXX-XXX |
| XX | XX | XX | XX | XX | XX | XX | XX | XX | | | n |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | Mean |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SD |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | | CV% |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SEM |
| XX | XX | XX | XX | XX | XX | XX | XX | XX | | | Minimum |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | Median |
| XX | XX | XX | XX | XX | XX | XX | XX | XX | | | Maximum |

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of 1 ng/mL are treated as 0 before the first quantifiable concentration and as missing elsewhere.

<sup>. =</sup> Value missing or not reportable.

### **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Subject number to be presented as follow: XXX-XXX
- Concentrations will be presented to same precision as in the bioanalytical data.
- Summary statistics presentation with respect to the precision of the bioanalytical data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

## Programmer Note:

• PK Time points are: predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose

Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables-sig.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_conc.sas DDMMYYYY HH:MM

# Tables 14.2.1.5 through 14.2.1.8 will be in the following format:

Table 14.2.1.5 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of 160 mg LOXO-292 Fasted (Treatment A) (Pharmacokinetic Population)

| | | eters ——— | Param | | | | | |
|---|---|---|---|---|---|---|---|---|
| parame | param5 | param4 | param3 | param2 | param1 | Study | Treatment | Subject |
| (units) | (units) | (units) | (units) | (units) | (units) | Period | Sequence | Number |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | X.XX | X | XXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXX | XXX-XXX |
| XX | XX | XX | XX | XX | XX | | | n |
| X.XXXX | XX.XX | XXX.X | XXX.X | X.XXX | XXX.X | | | Mean |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SD |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | CV% |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SEM |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | | | Minimum |
| X.XXXX | XX.XX | XXX.X | XXX.X | X.XXX | XX.XX | | | Median |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | | | Maximum |
| X.XXXX | XX.XX | XXX.X | XXX.X | X.XXX | XXX.X | | | Geom Mean |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | Geom CV% |

<sup>. =</sup> Value missing or not reportable.

Statistical Analysis Plan, 06 September 2018

#### **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Subject number to be presented as follow: XXX-XXX
- PK Parameters will be presented in the following order: AUC0-t <unit>, AUC0-inf <unit>, AUC%extrap <unit>, Cmax <unit>, Tmax <unit>, Kel <unit>, t1/2 <unit>, and CL/F <unit>
- n will be presented as an integer (with no decimal);
- Parameter values for exposure-based parameters (i.e. AUCs, AUC%extrap, Cmax, and CL/F) will be presented with, at maximum, the precision of the bioanalytical data, and, at minimum, 3 significant figures (to be determined by the PKist once the bioanalytical data are received).
  - Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2,
     Min and Max +0 with respect to the number of significant figures.
- Values for time-based parameters (i.e. Tmax, and t1/2) will be presented with 2 decimals.
  - Summary statistics for time-based parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of decimals.
- Values for rate constants (i.e. Kel) will be presented with 3 significant figures.
  - Summary statistics for Kel will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of significant figures.
- $\bullet$   $\,$  CV% and Geom CV% for all parameters will be presented with 1 decimal

Program: /CXXXXX/sas\_prg/pksas/pk-tables.sas DDMMYYYYY HH:MM
Program: /CXXXXX/sas\_prg/pksas/adam\_pkparam.sas DDMMYYYYY HH:MM

#### Table 14.2.1.9 will be in the following format:

Table 14.2.1.9 Intervals (Hours) Used for Determination of Plasma LOXO-292 Kel Values Following Administration of 160 mg LOXO-292 Fasted (Treatment A), Administration of 160 mg LOXO-292 Fed (Treatment B), Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fasted (Treatment C), and Coadministration of Multiple Dose Omeprazole + 160 mg LOXO-292 Fed (Treatment D) (Pharmacokinetic Population)

| Subject | Treatment | Trea | tment A | | | Treatment B | |
|---|---|---|---|---|---|---|---|
| Number | Sequence | Interval | R2 | n | Interval | R2 | n |
| XXX-XXX | XX | XX.X - XX.X | x.xxx | Х | XX.X - XX.X | x.xxx | X |
| XXX-XXX | XX | XX.X - XX.X | X.XXX | X | XX.X - XX.X | X.XXX | X |
| XXX-XXX | XX | XX.X - XX.X | X.XXX | X | XX.X - XX.X | X.XXX | Х |

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOKO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

R2 = Coefficient of determination

n = Number of points used in Kel calculation

<sup>. =</sup> Kel value not reportable.

## **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Interval start and stop times will be presented to 1 decimal or 3 significant figures minimum;
- R2 will be presented to 3 decimals;
- n will be presented as an integer (with no decimal)

## Per study design needs, the following changes are made to this table relative to Celerion standard:

1. Please add additional columns for Treatments C and D.

Program: /CXXXXX/sas\_png/pksas/kel-tables-xover.sas DDMMMYYYY HH:MM
Program: /CXXXXX/sas\_png/pksas/adam\_kel.sas DDMMMYYYY HH:MM

#### Tables 14.2.1.10 through 14.2.1.13 will be in the following format:

Table 14.2.1.10 Statistical Comparisons of Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of 160 mg LOXO-292 Fed (Treatment B)

Versus Administration of 160 mg LOXO-292 Fasted (Treatment A) (Pharmacokinetic Population)

| | | | Treatment<br>ometric I | _ | | Geometric<br>Mean | 90% | Intra-subject |
|---|---|---|---|---|---|---|---|---|
| Parameter | (unit) | В | (n) | A | (n) | Ratio | Confidence Intervals | CV% |
| Param1<br>Param2<br>Param3 | (unit)<br>(unit)<br>(unit) | X.XX<br>X.XX<br>X.XX | (n)<br>(n)<br>(n) | X.XX<br>X.XX<br>X.XX | (n)<br>(n)<br>(n) | X.XX<br>X.XX<br>X.XX | XX.XX - XXX.XX<br>XX.XX - XXX.XX<br>XX.XX - XXX.XX | X. XX<br>X. XX<br>X. XX |

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Parameters were ln-transformed prior to analysis.

Geometric least-squares means (LSMs) are calculated by exponentiating the LSMs from ANOVA.

Geometric Mean Ratio = 100\*(B/A)

Intra-subject CV% = 100 x (square root (exp[MSE]-1), where MSE = Residual variance from ANOVA.

## **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Geometric LSMs will be presented to same precision as Mean in the PK parameter table CPPar1,
- Geometric Mean Ratio, 90% CI and intra-subject CV% will be presented to 2 decimal places,
- PK parameters to be presented are AUC0-t, AUC0-inf, and Cmax

Program: /CXXXXX/sas\_prg/pksas/stats-tables-mixed.sas DDMMYYYYY HH:MM
Program: /CXXXXX/sas\_prg/pksas/adam\_statsmixed.sas DDMMYYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Table 14.3.1.1 Treatment-emergent Adverse Event Frequency by Treatment - Number of Subjects Reporting Events (% of Subject Dosed) (Safety Population)

| | | | | | Ί | reatmen | nt | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | | A | | В | OM | Æ Alone | 9 | С | | D | O | verall |
| Number of Subjects Dosed | Х | (100%) | Х | (100%) | Х | (100%) | Х | (100%) | Х | (100%) | X | (100%) |
| Number of Subjects with TE Adverse Events | X | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Number of Subjects without TE Adverse Events | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Nervous system disorders | X | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Dizziness | X | (XX%) | Х | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Headache | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Presyncope | X | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) | X | (XX%) |
| Respiratory, thoracic and mediastinal disorders | X | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Dry throat | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Oropharyngeal pain | X | (XX%) | X | (XX%) | X | (XX%) | X | (XX%) | X | (XX%) | X | (XX%) |
| Sinus congestion | X | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Sneezing | X | (XX%) | X | (XX%) | X | (XX%) | X | (XX%) | X | (XX%) | X | (XX%) |
| General disorders and administration site conditions | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Fatigue | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Thirst | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| etc. | | | | | | | | | | | | |

Note: \* Adverse events are classified according to the MedDRA Version 21.0 by System Organ Class and Preferred Term.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


TE = Treatment-emergent

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast.

Treatment OMP Alone: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Treatment C: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column. For each subject, please sort the AEs with same verbatim and preferred term by onset date/time. For any pair (e.g., AE\_S1, AE\_S2) of these AEs (for same subject, same verbatim and preferred term), if the onset date/time of AE\_S2 = resolved date/time of AE\_S1 and the grade of AE\_S2 < the grade level of AE\_S1, then mark the AE\_S2 with a flag like EVAUL\_FIG ="N". Then, for AE analysis (summary tables), please exclude the ones with EVAUL\_FIG ="N". Won't repeat this comment again.


Table 14.3.1.2 Treatment-emergent Adverse Event Frequency by Treatment - Number of Adverse Events (% of Total Adverse Events) (Safety Population)

| | | | | | 1 | reatmer | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| E Adverse Event* | | A | | В | Olv | 1P Alone | | С | Ι | ) | Overal | |
| Number of TE Adverse events | Х | (100%) | Х | (100%) | Х | (100%) | Х | (100%) | Х | (100%) | Х | <br>(100%) |
| Nervous system disorders | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| Dizziness | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Headache | X | (XX%) | Х | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Presyncope | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Respiratory, thoracic and mediastinal disorders | X | (XX%) | Χ | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Dry throat | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Oropharyngeal pain | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Sinus congestion | X | (XX%) | Х | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Sneezing | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| General disorders and administration site conditions | X | (XX%) | Х | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Fatigue | X | (XX%) | X | (XX%) | X | (XX%) | Х | (XX%) | X | (XX%) | X | (XX%) |
| Thirst | X | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | Х | (XX%) | X | (XX%) |
| etc. | | | | | | | | | | | | |

Note: \* Adverse events are classified according to the MedDRA Version 21.0 by System Organ Class and Preferred Term.

TE = Treatment-emergent

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

Treatment A: <description>
Treatment B: <description>

Treatment OMP Alone: <description>

Treatment C: <description>
Treatment D: <description>

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column.

Statistical Analysis Plan, 06 September 2018


Table 14.3.1.3 Treatment-Emergent Adverse Event Frequency by Treatment, Severity Grade, and Relationship to Study Drugs - Number of
Subjects Reporting Events (Safety Population)

| | T | Number of | | S | everit | ty Gra | de | Relationship to LOXO-292 | nip to LOXO-292 | Relationship to Omeprazole | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | Treat-<br>ment | Subjects with<br>Adverse Events | 1 | 2 | 3 | 4 | 5 | Related | Not Related | Related | Not Related |
| Dizziness | Α | X | X | X | X | X | X | X | X | X | X |
| Dry eye | В | X | X | X | X | X | X | X | X | X | X |
| Dry mouth | A | X | X | X | X | X | X | X | X | X | X |
| - | В | X | X | X | X | X | X | X | X | X | X |
| Dry throat | C | X | X | X | X | X | X | X | X | X | X |
| Ear pain | OMP Alone | X | X | X | X | X | X | X | X | X | X |
| Fatigue | D | X | X | X | X | X | X | X | X | X | X |
| Treatment A | | XX | X | Х | Х | X | x | X | Х | X | X |
| Treatment B | | XX | X | X | X | X | X | X | X | X | X |
| Treatment OMP Alor | ne | XX | X | X | X | X | X | X | X | X | X |
| Treatment C | | XX | X | X | X | X | X | X | X | X | X |
| Treatment D | | XX | X | X | X | X | X | X | X | X | X |
| Overall | | XX | X | X | X | X | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 21.0 by System Organ Class and Preferred Term.

TE = Treatment-emergent; AE = Adverse event

Severity Grade: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately lifethreatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection. If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

When a subject experienced the same TEAE at more than one level of severity during a treatment period, only the most severe one was counted.

When a subject experienced the same TEAE at more than one level of drug relationship during a treatment period, only the one related to study drugs was counted.

Treatment A: <description>

Treatment B: <description>

Treatment OMP Alone: <description>

Treatment C: <description>
Treatment D: <description>

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Table 14.3.1.4 Treatment-Emergent Adverse Event Frequency by Treatment, Severity Grade, and Relationship to Study Drugs - Number of Adverse Events (Safety Population)

| Treat- | | Number of | | S | everi | ty Grad | de | Relationsh | ip to LOXO-292 | Relationsh | nip to Omeprazole |
|---|---|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | | Adverse Events | 1 | 2 | 3 | 4 | 5 | Related | Not Related | Related | Not Related |
| Dizziness | Α | X | Х | X | X | X | X | X | X | Х | X |
| Dry eye | В | X | X | X | X | X | X | X | X | X | X |
| Dry mouth | A | X | X | X | X | X | X | X | X | X | X |
| | В | X | X | X | X | X | X | X | X | X | X |
| Dry throat | C | X | X | X | X | X | X | X | X | X | X |
| Ear pain | OMP Alone | Y X | X | X | X | X | X | X | X | X | X |
| Fatigue | D | X | X | X | X | X | X | X | X | X | X |
| Treatment A | | XX | X | X | X | X | X | X | X | X | X |
| Treatment B | | XX | X | X | X | X | X | X | X | X | X |
| Treatment OMP Alor | ne | XX | X | X | X | X | X | X | X | X | X |
| Treatment C | | XX | X | X | X | X | X | X | X | X | X |
| Treatment D | | XX | X | X | X | X | X | X | X | X | X |
| Overall | | XX | X | X | X | X | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 21.0 by System Organ Class and Preferred Term.

TE = Treatment-emergent; AE = Adverse event

Severity Grade: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-

threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection. If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

Treatment A: <description>
Treatment B: <description>

Treatment OMP Alone: <description>

Treatment C: <description>
Treatment D: <description>

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Page X of X

#### Table 14.3.2.1 Serious Adverse Events (Safety Population)

| Subject | Treat- | | Adverse | PT*/ | On | set/Resolut<br> | ion | | Severity | | | Action for LOXO-292/ | Relationship to LOXO-292/ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | ment | TE?^ | Event | SOC | Day | Date | Time | Freq* | Grade | Ser* | Outcome | Omeprazole | Omeprazole |
| XXX-XXX | Х | Yes | XXXXXXXXXX | XXXXXXX/<br>XXXXXXXX | XX/<br>XX | DDMMYYYY/<br>DDMMYYYYY | | Inter. | XXXXXX | NS | Resolved | XXXXXXXXXX/<br>XXXXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXXX |

Note: \* Adverse events are classified according to MedDRA Version 21.0 by System Organ Class and Preferred Term.

TE = Treatment-emergent; PT = Preferred Term; SOC = System Organ Class, Onset day is relative to Period 1 Day 1.

Freq\* represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous

Ser\* represents Serious: NS = Not Serious

Severity Grade: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately

life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection.

Treatment A: <description>

Treatment B: <description>

Treatment OMP Alone: <description>

Treatment C: <description>

Treatment D: <description>

Program: /CAXXXXX/sas\_prq/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: if there are no serious adverse events reported, there will be just one table (Table 14.3.2.1) with the statement "There was no serious adverse event recorded during the study."

Statistical Analysis Plan, 06 September 2018


Tables 14.3.4.2-14.3.4.4 will have the following format.

Page 1 of X Table 14.3.4.1 Out-of-Range Values and Recheck Results - Serum Chemistry (Safety Population)

| Subject<br>Number | Age\$/<br>Sex | Study<br>Period | Treatment | Day | Hour | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XX/M | Screen<br>X | Х | -x<br>x | -XX.XX<br>XX.XX | DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY | XX HN G1<br>XX<br>XX LY- | XX<br>XX<br>XX LN | XX<br>XX<br>XX | XX LY- | XX HN<br>XX<br>XX |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Arrange alphabetically by lab test name.

Note: \$ Age is calculated from the date of first dosing

Abnormal flag: H = Above Reference Range, L = Below Reference Range

Computer Clinical significance: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

Treatment A: <description>

Treatment B: <description>

Treatment C: <description>

Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

| Subject<br>Number | | | Treatment | Day | Hour | Date | Time | Department | Test | Result | Reference Range | Unit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XX/X | X | X | -X | -x.xx | DDMMMYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX | X - X | mg/dL |
| | | | | | | | | Serum Chemistry | | XXX HYR+G | 3 X - X | mg/dL |
| | | | | X | XX.XX | DD <b>MM</b> MYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HY- G | 2 X - X | mg/dL |
| | | | | X | XX.XX | DDMMMYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HN G | X – X | ma/dT |

Programmer Note: All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table.

If there were no CS values as deemed by PI (i.e., no "CS" or "Clinically Significant" in the PI flag or comment field in the laboratory dataset), then this table will contain only the statement: "There were no laboratory values deemed clinically significant by the PI in the study."

Note: \$ Age is calculated from the date of first dosing

H = Above Reference Range, L = Below Reference Range

Computer: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

Treatment A: <description>
Treatment B: <description>
Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program : /CAXXXXX/ECR/sas\_prg/stsas/tab/PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


#### Tables 14.3.5.1, 14.3.5.3, and 14.3.5.5 will have the following format.

Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline - Serum Chemistry (Safety Population)

| | | Time | ime - | | Treatment | | | | Change From Baseline | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test (unit) | Normal Range# | Point | Statistic | Α | В | С | D | A | В | С | D |
| Parameter1 (unit) | XX - XX | Baseline | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | | | | |
| | | Day 4 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX |
| | | Day 7/8\$ | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX |

<Programmer note: Similar for remaining laboratory tests. Sort alphabetically by lab test name.>

Note: # Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

Baseline is Day -1 of Period 1 and Day 7 of previous period for Period 2, 3, 4 and is the last non-missing predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments. Day 7 measurement of Period 1, 2, 3 was used twice as postdose value of Period 1, 2, 3 and baseline value of Period 2, 3, 4.

Treatment A: <description>

Treatment B: <description>

Treatment C: <description>

Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


<sup>\$</sup> Day 7 for Period 1, 2, 3 and Day 8 for Period 4

#### Tables 14.3.5.2, 14.3.5.4, and 14.3.5.6 will have the following format.


| | | | | Bas | eline | L | | Bas | eline | N | Bas | eline | e H |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Po | stdos | e | | Po | stdos | е | Pos | tdose | 9 |
| Laboratory<br>Test (units) | Treat-<br>mend | Time<br>Point | | L | N | Н | | L | N | Н | L | N | Н |
| Testname (unit) | | Day 4 | | Х | XX | Х | | | XX | X | Х | XX | Х |
| | | Day 7 | | X | XX | Х | | X | XX | X | Х | XX | Х |
| | В | Day 4 | | X | XX | Х | | X | XX | X | Х | XX | Х |
| | | Day 7 | | X | XX | Х | | Х | XX | X | Х | XX | X |
| | C | Day 4 | | X | XX | Х | | Х | XX | X | Х | XX | Х |
| | | Day 7/8 | \$ | X | XX | X | | Х | XX | X | X | XX | Х |
| | D | Day 4 | | X | XX | Х | | Х | XX | X | Х | XX | X |
| | | Day 7/8 | \$ | X | XX | Х | | Х | XX | X | Х | XX | Х |
| < > | < > | romaini | na lah | t . | ~·· + o | ata II | 70 M | TAT | i+bin | Movmol | Dange | _ | O |

<Programmer note: Similar for remaining laboratory tests. Use N = Within Normal Range, O = Outside Normal Range for urinalysis shift table.>

Note: N = Within Normal Range, L = Below Normal Range, H= Above Normal Range.

\$ Day 7 for Period 3 and Day 8 for Period 4

Baseline is Day -1 of Period 1 and Day 7 of previous period for Period 2, 3, 4 and is the last non-missing predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments. Day 7 measurement of Period 1, 2, 3 was used twice as postdose value of Period 1, 2, 3 and baseline value of Period 2, 3, 4.

Table 14.3.5.2 Clinical Laboratory Shift from Baseline - Serum Chemistry (Safety Population)

Treatment A: <description>

Treatment B: <description>

Treatment C: <description>

Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/tab\_programname.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Table 14.3.5.7 Vital Sign Summary and Change from Baseline (Safety Population)

| Witel Cim | T-1 | | | Tı | eatmen | t | C | hange From | n Baseline | e |
|---|---|---|---|---|---|---|---|---|---|---|
| Vital Sign<br>Parameter (unit) | Time<br>Point | Statistic | Α | В | С | D | A | В | С | D |
| Parameter1 (unit) | Day -1/1\$ | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | | | | |
| | Postdose Hour 2 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX |
| | Postdose Hour 72 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>XX.X<br>XX.X<br>XX.XX | X.XXX<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX |

<Programmer note: Similar for remaining vital sign parameters. Treatment D has an additional time point: Postdose Hour
168.>

Note: \$ Day -1 for Period 1 and Day 1 for Period 2, 3, 4

Baseline is Day -1 of Period 1 and Day 1 predose of Period 2, 3, 4 and is the last non-missing predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments.

Treatment A: <description>
Treatment B: <description>
Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Page 1 of X Table 14.3.5.8 12-Lead Electrocardiogram Summary and Change from Baseline (Safety Population)

| RGG | Time | | Treatment Change From Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ECG<br>Parameter (unit) | Point | Statistic | Α | В | С | D | A | В | С | D |
| Parameter1 (unit) | Day -1/1\$ | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX | XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | | | | |
| | Postdose Hour 2 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>XX.X<br>XX.X<br>XX.XX | XX.X | XX<br>XX.XX<br>X.XXX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX |
| | Postdose Hour 72 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX |

<Programmer note: Similar for remaining ECG parameters. Treatment D has an additional time point: Postdose Hour 168.>

Note: \$ Day -1 for Period 1 and Day 1 for Period 2, 3, 4

Baseline is Day -1 of Period 1 and Day 1 predose of Period 2, 3, 4 and is the last non-missing

predose measurement prior to dosing of LOXO-292, including rechecks and unscheduled assessments.

Treatment A: <description>
Treatment B: <description>
Treatment C: <description>

Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


#### 11. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final CSR. These listings will be generated from the Celerion SDTM Tabulation Model 1.4 mapped in accordance with SDTM Implementation Guide 3.2. All listings will be presented in Courier New size font 9.

Statistical Analysis Plan, 06 September 2018


Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Laboratory Group | Test Name | Sex | Age Category | Normal Range | Unit |
|------------------|-----------|--------|--------------|--------------|-------|
| Serum Chemistry | Test Name | XXXXXX | XX | XX - XX | units |
| _ | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| Hematology | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |

<Programmer note: Sort alphabetically by lab test name within each lab group.>

<similar for remaining Laboratory Groups and Test Names>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Appendix 16.2.1 Subject Discontinuation (Safety Population)

| Subject<br>Number | Treatment<br>Sequence | Study<br>Period | Date | Completed Study? | Primary | Discontinuation | Reason |
|---|---|---|---|---|---|---|---|
| XXX-XXX | ABCD | Post | DDMMYYYY | YES | | | |
| XXX-XXX | ABCD | Post | DDMMMYYYY | YES | | | |
| XXX-XXX | ABCD | Post | DDMMMYYYY | YES | | | |
| XXX-XXX | ABCD | Post | DDMMMYYYYY | YES | | | |
| XXX-XXX | ABCD | Post | DD <b>MM</b> MYYYY | NO | Adverse | Event | |
| XXX-XXX | ABCD | Post | DD <b>MM</b> MYYYY | YES | | | |
| XXX-XXX | ABCD | Post | DD <b>MM</b> MYYYY | YES | | | |
| XXX-XXX | ABCD | Post | DD <b>MM</b> MYYYY | YES | | | |

Note: Treatment A: 160 mg LOXO-292 (2 x 80 mg capsules) at Hour 0 on Day 1 administered under fasting conditions.

Treatment B: 160 mg LOXO-292 (2  $\times$  80 mg capsules) at Hour 0 on Day 1 administered 30 minutes after the start of a high fat breakfast. Treatment C: Multiple daily doses of 40 mg omeprazole (1  $\times$  40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2  $\times$  80 mg capsules) coadministered at Hour 0 on Day 1 under fasting conditions.

Treatment D: Multiple daily doses of 40 mg comeprazole (1 x 40 mg capsule) from Day 1 to Day 7 with 160 mg LOXO-292 (2 x 80 mg capsules) coadministered at Hour 0 on Day 1, 30 minutes after the start of a high fat breakfast.

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Appendix 16.2.4.1 Demographics (Safety Population)

| Subject<br>Number | Date of<br>Birth | Age*<br>(yr) | Sex | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | Body Mass<br>Index<br>(kg/m^2) | Informed<br>Consent<br>Date | Informed<br>Consent<br>Version Date |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | DD <b>MM</b> YYYY | XX | AAAAAA | AAAAAAA | АААААААА | XXX | XX.XX | XX.XX | DDMMMYYYY | DD <b>MM</b> MYYYY |
| XXX-XXX | DD <b>MM</b> YYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DD <b>MM</b> MYYYY | DD <b>MM</b> YYYYY |
| XXX-XXX | DD <b>MM</b> YYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DD <b>MM</b> MYYYY | DD <b>MM</b> YYYYY |
| XXX-XXX | DD <b>MM</b> YYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYYY |
| XXX-XXX | DD <b>MM</b> YYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYYY |
| XXX-XXX | DD <b>MM</b> YYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYYY |
| XXX-XXX | DD <b>MM</b> YYYY | XX | AAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYY |

Note: \* Age is calculated form the date of first dosing.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Appendix 16.2.4.2 Updated Informed Consent (Safety Population)

| Subject<br>Number | Date Subject Signed<br>Informed Re-Consent | Informed Re-Consent<br>Version Date | Reason for<br>Re-Consent |
|---|---|---|---|
| XXX-XXX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYY | XXXXXXXXXXXX |
| XXX-XXX | DDMMYYYYY | DDMMYYYYY | XXXXXXXXXXXXXXX |
| XXX-XXX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYY | XXXXXXXXXXXXXX |
| XXX-XXX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYY | XXXXXXXXXXXXXX |
| XXX-XXX | DDMMYYYYY | DD <b>MM</b> YYYY | XXXXXXXXXXXXXX |
| XXX-XXX | DDMMYYYYY | DDMMYYYYY | XXXXXXXXXXXXXXX |
| XXX-XXX | DDMMYYYYY | DDMMYYYYY | XXXXXXXXXXXXXXX |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

## Loxo Oncology, Inc. LOXO-292, LOXO-RET-18015

# Celerion, Clinical Study Report No. CA24336

Appendix 16.2.4.3 Physical Examination (Safety Population)

| | Treatment<br>Sequence | Period | Day Hour | Date | Body<br>System | Answer or<br>Result | Comment |
|---|---|---|---|---|---|---|---|
| xxx-xxx | ABCD | Screen | | DDMMYYYY | Was PE performed?<br>General<br>HEENT<br>< > | Yes<br>Normal<br>Normal<br>< > | |
| | | 1 | -1 Check-in | DDMMYYYY | Was PE performed?<br>HEENT<br>< > | Yes<br>Unchanged<br>< > | |

Note: Treatment A: <description>
Treatment B: <description>
Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM


# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18015

Celerion, Clinical Study Report No. CA24336


Appendix 16.2.4.4 Medical and Surgical History (Safety Population)

| | | | Date | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Any<br>History? | Study<br>Period | Category | Body system | Start | End | Ongoing? | Condition or Events |
| XXX-XXX | XXX | Screen | Medical<br>Surgical | XXXXXXXXXX | DDMMYYYY<br>DDMMYYYYY | DD <b>MM</b> YYYY<br>DD <b>MM</b> YYYY | YES | XXXXXXX XXXXXX XXXXXXXX |
| XXX-XXX | XXX | Screen | Medical | XXXXXXXXXX | DD <b>MM</b> YYYY | DD <b>MM</b> YYYY | NO | |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM
Celerion, Clinical Study Report No. CA24336


Appendix 16.2.4.5 Nicotine Use (Safety Population)

| Subject<br>Number | | Substance | Description of Use | Start<br>Date | End<br>Date |
|---|---|---|---|---|---|
| XXX-XXX | Screen | XXXXXXXX XXX | XXXXX XXXXXXX XXXXXX | DDMMYYYY | DD <b>MM</b> MYYYY |


Appendix 16.2.5.1.1 Inclusion Criteria

| 1. | Healthy, | adult, | male or | female | (of | non-childbearing | potential | only), | 18-55 | years | of | age, | inclusive, | at | screening. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | | | | | | _ | - | 4., | | - | | | | | _ |

2. <> 3. <> 4. <> 5. <>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


### Celerion, Clinical Study Report No. CA24336


#### Appendix 16.2.5.1.2 Exclusion Criteria

- 1. Is mentally of legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
- 3. <>
- 4. <> 5. <> 6. <>
- 7. <>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Appendix 16.2.5.2 Subject Eligibility (Safety Population)


| Subject<br>Number | Study<br>Period | Did subject meet all eligibility criteria? | Specify |
|---|---|---|---|
| XXX-XXX | Screen | YES | |
| XXX-XXX | Screen | NO | <pre><this column="" data="" if="" is="" only="" present="" presented=""></this></pre> |


Appendix 16.2.5.3.1 Check-in Criteria

- Did the Subject report any study restriction violations since the last study visit?
   IF YES TO ANY QUESTION, WAS SUBJECT APPROVED FOR STUDY?

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


### Celerion, Clinical Study Report No. CA24336


#### Appendix 16.2.5.3.2 Check-in Responses (Safety Population)

| Subject | Treatment | Study | | Check-in Criteria | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Sequence | | Day | Hour | Date | Time | X | Х | Specify |
| XXX-XXX | ABCD | 1 | Х | Check-in | DDMMYYYYY | hh:mm:ss | YES | YES | <pre><this column="" data="" if="" is="" only="" present="" prints=""></this></pre> |

Note: Treatment A: <description>

Treatment B: <description>

Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Celerion, Clinical Study Report No. CA24336


#### Appendix 16.2.5.4.1 Test Compound Description

| Compound | Form | Route |
|-----------------|------|-------|
| XXXXXXXXXXXXXXX | < > | XXXX |
| XXXXXXXXXXXXX | < > | XXXX |

Celerion, Clinical Study Report No. CA24336


Appendix 16.2.5.4.2 Test Compound Administration Times (Safety Population)

| Subject<br>Number | _ | Treatment | Day | Hour | Date | Actual<br>Time | Compound | Dosage | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | 1 2 | X<br>X | X<br>X | 0 | DD <b>MM</b> YYYY<br>DDMMYYYY | | XXXXXXXXXX | < ><br>< > | <pre><this column="" data="" if="" is="" only="" present="" prints=""></this></pre> |

Note: Treatment A: <description>

Treatment B: <description>
Treatment C: <description>

Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Celerion, Clinical Study Report No. CA24336


Appendix 16.2.5.5 PK Blood Draw Times (Safety Population)

| Subject<br>Number | _ | Treatment | Day | Hour | Date | Actual<br>Time | Bioassay | Comments |
|---|---|---|---|---|---|---|---|---|
| XXX-XXX | 1 | X | 1 | -X.XX | DDMMYYYY | X:XX:XX | XXXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> MYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> YYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> YYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> MYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> MYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> MYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> YYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> MYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | 2 | XX.XX | DD <b>MM</b> MYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> YYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DD <b>MM</b> YYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | 3 | XX.XX | DD <b>MM</b> YYYYY | X:XX:XX | XXXXXXXXXX | |

Note: Treatment A: <description>

Treatment B: <description> Treatment C: <description>

Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule)

from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM


Statistical Analysis Plan, 06 September 2018


Appendix 16.2.5.6 Phone Call (Safety Population)

| _ | 4 | Was a Teleph<br>Performed? | Day | Date | Time | If No, Reason* |
|---|---|---|---|---|---|---|
| XXX-XXX | 4 | YES | <br>XX | DDMMYYYY | HH:MM | XXXXXXXXXXXXX |

Note: \* Reason options: 3 call attempts with no subject return call; Phone Disconnected; Wrong Number


Appendix 16.2.5.7 Meal Times (Safety Population)

| Subject<br>Number | Study<br>Period Treatment | | Day | Hour | Event | Date | Start<br>Time | | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | | | x<br>x | -XX.XX<br>XX.XX<br>-XX.XX<br>-XX.XX<br>XX.XX<br>-XX.XX<br>-XX.XX | DINNER SNACK LUNCH DINNER SNACK BREAKFAST LUNCH DINNER | DINNER DDMMYYYY SNACK DDMMYYYY JUNCH DDMMYYYY DINNER DDMMYYYY SNACK DDMMYYYY SREAKFAST DDMMYYYY JUNCH DDMMYYYY | | XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX: | |
| | 2 | В | х | -XX.XX<br>-XX.XX<br>-XX.XX<br>XX.XX<br>-XX.XX<br>-XX.XX<br>-XX.XX<br>-XX.XX<br>-XX.XX | DINNER<br>SNACK<br>BREAKFAST<br>LUNCH<br>DINNER<br>SNACK<br>BREAKFAST | DDMMYYYYY<br>DDMMYYYYY<br>DDMMYYYYY<br>DDMMYYYYY<br>DDMMYYYYY | XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX | XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX<br>XX:XX: | |

Note: Treatment A: <description>
Treatment B: <description>
Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

### Celerion, Clinical Study Report No. CA24336


#### Appendix 16.2.5.8 Prior and Concomitant Medications (Safety Population)

| Subject Treat-<br>Number ment | - | Prior to<br>Study? | Medication<br>(WHO* Term) | Dosage | Route | Frequency | Start<br>Day/Date/Time | Stop<br>Day/Date/Time | | | Continuing |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX X | No<br>Yes | Yes | None<br>ACETAMINOPHEN<br>(ACETAMINOPHEN | _ | BY MOUTH | AS NEEDED | XX/DDMMYYYY/<br>HH:MM | XX/DDMMYYYY/<br>HH:MM | XXXXX | XXX | YES |

Note: \* Concomitant medications are coded with WHO Dictionary Version Mar2017 B3.

^ Med = Medication; UNK = Unknown

Prior medication was medication taken prior to study drug administration.

Start and stop day is relative to Period 1 Day 1.

Treatment A: <description>
Treatment B: <description>

Treatment OMP Alone: <description>

Treatment C: <description>
Treatment D: <description>

### Celerion, Clinical Study Report No. CA24336


#### Appendix 16.2.7.1 Adverse Events (I of II) (Safety Population)

| | | | 7.1 | Time from<br>Last Dose | se Onset | | | | Resolved | Duration | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Treatment | TE?^ | Adverse Event/<br>Preferred Term* | (DD:HH:MM) | Day | Date | Time | Day | Date | Time | (DD:HH:MM) |
| XXX-XXX | | None | | | | | | | | | |
| XXX-XXX | Х | Yes | XXXXXXXXXXXXX/<br>XXXXXXXXXXX | XX:XX:XX | XX | DD <b>MM</b> YYYY | X:XX | XX | DD <b>MM</b> YYYY | X:XX | XX:XX:XX |
| | | No | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXX | XX:XX:XX | XX | DD <b>MM</b> MYYYY | X:XX | XX | DDMMYYYY | X:XX | XX:XX:XX |

Note: \* Adverse events are classified according to MedDRA Version 21.0 by System Organ Class and Preferred Term.

^ TE = Treatment-emergent, Onset and resolved day is relative to Period 1 Day 1.

Treatment A: <description>
Treatment B: <description>
Treatment OMP Alone: <description>
Treatment C: <description>

Treatment C: <description>
Treatment D: <description>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


#### Appendix 16.2.7.2 Adverse Events (II of II) (Safety Population)

| Subject | Treat- | - Adverse | | Onset | | | | | | Action for<br>LOXO-292/ | | Other<br>Action | Relationship to |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | ment | Event | Day | Date | Time | Freq* | Severity | Ser* | Outcome | | • | Taken | Omeprazole |
| XXX-XXX | | None | | | | | | | | | | | |
| XXX-XXX | X | XXXXXXX | XX | DD <b>MM</b> YYYY | XX:XX | Inter. | Grade 1 | NS | Resolved | | Changed/<br>Changed | | Not Related to |

Note: Ser\* represents Serious: NS = Not Serious

Freq\* represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous

Onset day is relative to Period 1 Day 1.

Severity/Intensity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately

life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection.

Treatment A: <description>
Treatment B: <description>

Treatment OMP Alone: <description>

Treatment C: <description>
Treatment D: <description>

\_

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Appendix 16.2.7.3 Adverse Event Non-Drug Therapy (Safety Population)

| | | | | Onset | | | Resolved | | Therapy | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | | Adverse | | | | | | | | | |
| Number | Treatment | Event | Day | Date | Time | Day | Date | Time | Date | Time | Description |
| XXX-XXX | X | DRY LTPS | XX | DDMMMYYYY | X · XX | XX | DDMMMYYYY | X:XX | DDMMMYYYY | XX • XX | PETROLEUM JELLY |

Note: Onset and resolved day is relative to Period 1 Day 1.

Treatment A: <description>
Treatment B: <description>

Treatment OMP Alone: <description>

Treatment C: <description>
Treatment D: <description>


#### Appendix 16.2.7.4 Adverse Event Preferred Term Classification (Safety Population)

| | | | | | | Onset | |
|---|---|---|---|---|---|---|---|
| Subject | | Adverse | | | | | |
| Number | Treatment | Event | Preferred Term* | Body System | Day | Date | Time |
| XXX-XXX | X | XXXXXXX XXXXX XXXXX XXXXXX | XXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX | DDMMYYYYY | X:XX |

Note: \* Adverse events are classified to MedDRA Version 21.0 by System Organ Class and Preferred Term.

Onset day is relative to Period 1 Day 1.

Treatment A: <description>
Treatment B: <description>
Treatment OMP Alone: <description>

Treatment C: <description>

Treatment D: <description>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


#### Appendices 16.2.8.1.2-16.2.8.1.4 will have the following format.

Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)

| Subject<br>Number | Age\$/<br>Sex | Study<br>Period | Treatment | Day | Hour | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XX/M | Screen<br>X | х | -X<br>X | -XX.XX<br>XX.XX | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XX HN<br>XX<br>XX LY- | XX<br>XX<br>XX I.N | XX<br>XX<br>XX | XX<br>XX<br>XX L.Y- | XX HN<br>XX<br>XX |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Arrange alphabetically by lab test name.

```
Note: $ Age is calculated from the date of first dosing.

H = Above Reference Range, L = Below Reference Range

Computer Clinical Significance: N = Not Clinically Significant, Y = Clinically Significant
```

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event

Treatment A: <description>
Treatment B: <description>
Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


#### Celerion, Clinical Study Report No. CA24336


Appendix 16.2.8.1.5 Clinical Laboratory Report - Comments (Safety Population)

| Subject<br>Number | | Treatment | Day | Hour | Date | Department | Test | Result | Unit | Comment |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | X | Х | -X | -X.X | DD <b>MM</b> MYYYY | Other Tests | Fibrinogen | XXX | | Not significant in the context of this study. |

Note: Treatment A: <description>

Treatment B: <description>
Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg cmeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Celerion, Clinical Study Report No. CA24336

Appendix 16.2.8.2 Vital Signs (Safety Population)

| Cubicat | C+ndr | | | | | | | | Pressure | | Pulse | Respir-<br>ation | - Temper- | Weight | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Study<br>Period | Treatmen | t Day | Hour | Date | Time | | | Systolic/ | | | (rpm) | ature<br>(°C) | (kg) | Comments |
| XXX-XXX | Screen | | | | DDMMYYYY | X:XX:XX | | | | | | | | XXX.X | |
| | | | | | DD <b>MM</b> MYYYY | X:XX:XX | SITX | Right | XXX/ | XX | XX | XX | XX.X | | |
| | 1 | X | -X | -XX.X | DDMMYYYYY | XX:XX:XX | | | | | | | | XXX.X | |
| | | | X | -X.X | DD <b>MM</b> YYYYY | X:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |
| | | | | X.X | DDMMYYYYY | X:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |
| | 2 | X | X | -x.x | DDMMYYYYY | X:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |
| | | | | X.X | DDMMYYYYY | X:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |
| | | | | R | DDMMYYYYY | XX:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |
| | | | X | -X.X | DD <b>MM</b> YYYYY | X:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |
| | | | | X.X | DD <b>MM</b> YYYYY | X:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |
| | | | X | XX.X | DDMMYYYYY | XX:XX:XX | SITX | Right | XXX/ | XX | XX | XX | | | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Note: SITX = X-minute sitting, R = Recheck Value.

Treatment A: <description>
Treatment B: <description>
Treatment C: <description>
Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg cmeprazole (1 x 40 mg capsule) from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| Subject<br>Number | Study<br>Period | Treatment | Day | Hour | Date | Time | Result | Heart<br>Rate<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF*<br>(msec) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | Screen | | | | DD <b>MM</b> YYYY | X:XX:XX | Normal | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | 1 | X | X | -x.xx | DDMMYYYYY | X:XX:XX | ANCS | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | | X.XX | DD <b>MM</b> YYYYY | X:XX:XX | Normal | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | 2 | X | X | -x.xx | DD <b>MM</b> YYYYY | X:XX:XX | ANCS | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | | X.XX | DDMMYYYYY | X:XX:XX | Normal | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | X | -x.xx | DDMMYYYYY | X:XX:XX | Normal | XX | XXX.X | XX.X | XXX.X | XXX.X # | |
| | | | | X.XX | DDMMYYYYY | X:XX:XX | Normal | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | X | X.XX | DD <b>MM</b> YYYYY | X:XX:XX | Normal | XX | XXX.X | XX.X | XXX.X | XXX.X @ | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Note: ANCS = Abnormal, Not Clinically Significant

QTcF\* = QT corrected for heart rate using Fridericia's correction. # = QTc > 450, @ = QTc change from baseline greater than 30 msec

Treatment A: <description> Treatment B: <description> Treatment C: <description> Treatment D: <description>

Prior to Treatment C or D at Period 3, subjects were administered with multiple daily doses of 40 mg omeprazole (1 x 40 mg capsule)

from Day -4 to Day -1 of Period 3.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYYY HH:MM

Statistical Analysis Plan, 06 September 2018


# 16.1.9.2 Statistical Outputs























